CLINICAL TRIAL: NCT06364917
Title: DISCERN: Dual Immune Strategy Versus Single Checkpoint Inhibition Efficacy Response in PDL-1 Negative Non-Small Cell Lung Cancer (NSCLC)
Brief Title: DISCERN: Dual Versus Single ICB in PDL-1 Negative NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Aakash Desai, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012781 (UAB2432); Robert Award (Other: The University of Alabama at Birmingham)
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Paclitaxel; Pemetrexed; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- single agent immune checkpoint blockade (ICB) + chemotherapy (CT) (Experimental): 200 mg of Pembrolizumab will be administered intravenously (IV) every 3 weeks (Q3W) for 4 cycles.
  Combination chemotherapy:
  For squamous NSCLC: Carboplatin (dose according to area under the curve (AUC) 6) + paclitaxel 200 mg/m².
  For non-squamous NSCLC: Carboplatin (AUC 5) + pemetrexed 500 mg/m². Maintenance Therapy for Non-Squamous NSCLC: Pembrolizumab 200 mg + pemetrexed 500 mg/m² Q3W for up to 2 years.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed
- dual agent immune checkpoint blockade (ICB) + chemotherapy (CT) (Experimental): Drug 1: 360 mg of Nivolumab will be administered intravenously (IV) every 3 weeks (Q3W).
  Drug 2: 1 mg/kg of Ipilimumab will be administered intravenously (IV) every 6 weeks (Q6W) for 2 cycles.
  Combination Chemotherapy:
  For squamous NSCLC: Carboplatin (AUC 6) + paclitaxel 200 mg/m². For non-squamous NSCLC: Carboplatin (AUC 5) + pemetrexed 500 mg/m². Maintenance Therapy for Non-Squamous NSCLC: Nivolumab 360 mg Q3W + Ipilimumab 1mg/kg Q6W for up to 2 years.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Pembrolizumab — The dosing regimens for Pembrolizumab (200 mg Q3W), are based on established FDA-approved dosages for the treatment of NSCLC, ensuring a balance between efficacy and tolerability. These doses are selected based on extensive clinical experience indicating optimal response rates with manageable safety profiles in the target population. The route of administration (intravenous) is chosen for its direct delivery into the bloodstream, ensuring maximum bioavailability and consistency of dosing.
  Arms: single agent immune checkpoint blockade (ICB) + chemotherapy (CT)
Drug: Carboplatin — The combination therapy dosages for Carboplatin are aligned with standard chemotherapy protocols for NSCLC, tailored to minimize toxicity while maintaining therapeutic efficacy. This dosing strategy is justified by previous phase 3 trials demonstrating the effectiveness and safety of these regimens in advanced NSCLC patients.
Drug: Paclitaxel — The combination therapy dosages for Paclitaxel are aligned with standard chemotherapy protocols for NSCLC, tailored to minimize toxicity while maintaining therapeutic efficacy. This dosing strategy is justified by previous phase 3 trials demonstrating the effectiveness and safety of these regimens in advanced NSCLC patients.
Drug: Pemetrexed — The combination therapy dosages for Pemetrexed are aligned with standard chemotherapy protocols for NSCLC, tailored to minimize toxicity while maintaining therapeutic efficacy. This dosing strategy is justified by previous phase 3 trials demonstrating the effectiveness and safety of these regimens in advanced NSCLC patients.
Drug: Nivolumab — The dosing regimens for Nivolumab (360 mg Q3W) are based on established FDA-approved dosages for the treatment of NSCLC, ensuring a balance between efficacy and tolerability. These doses are selected based on extensive clinical experience indicating optimal response rates with manageable safety profiles in the target population. The route of administration (intravenous) is chosen for its direct delivery into the bloodstream, ensuring maximum bioavailability and consistency of dosing.
  Arms: dual agent immune checkpoint blockade (ICB) + chemotherapy (CT)
Drug: Ipilimumab — The dosing regimens for Ipilimumab (1 mg/kg Q6W) are based on established FDA-approved dosages for the treatment of NSCLC, ensuring a balance between efficacy and tolerability. These doses are selected based on extensive clinical experience indicating optimal response rates with manageable safety profiles in the target population. The route of administration (intravenous) is chosen for its direct delivery into the bloodstream, ensuring maximum bioavailability and consistency of dosing.
  Arms: dual agent immune checkpoint blockade (ICB) + chemotherapy (CT)

SUMMARY:
The purpose of this study, known as DISCERN, is to compare two different treatments for a type of lung cancer called non-small cell lung cancer (NSCLC) that does not show a marker known as PD-L1. This study will help us understand if using two types of immune therapy together with chemotherapy is better than using one type of immune therapy with chemotherapy. We're doing this by looking at changes in the subject's cancer's DNA in the blood after starting treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female aged 18 years or older.
4. Participants must have histologically or cytologically confirmed non-small cell lung cancer which is stage IV
5. Participants should not have a known sensitizing mutation for which an FDA-approved.

   targeted therapy for NSCLC exists in first line (e.g., EGFR, ALK, ROS1, BRAF, RET, NTRK, and MET sensitizing mutations
6. Participants should not have received prior systemic anticancer therapy for advanced or metastatic disease. For patients who are recently diagnosed and received one cycle of chemotherapy while awaiting NGS/PDL-1 testing are allowed on study after discussion with medical monitor.
7. Participants should have measurable disease based on RECIST 1.1 as determined by the local site investigator/radiology assessment. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. Participants should have a life expectancy of at least 3 months.
9. Participants should have a performance status of 0, 1 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
10. Participants should have provided tumor tissue from locations not radiated prior to biopsy; fresh formalin fixed specimens or archival samples which have been determined as PD-L1 status <1% or negative prior to randomization.
11. Participants should have been evaluated for circulating tumor DNA at baseline which has been determined to be detected, present or positive.
12. Participants with CNS metastases are eligible if all metastases have been treated and have remained stable without growth for at least 2 weeks post-treatment, the participant's neurological status has returned to baseline or remained stable for at least 2 weeks, and any use of corticosteroids for CNS metastases is at a dose of ≤10 mg daily prednisone (or an equivalent dose of another corticosteroid) and has been stable for at least 2 weeks before enrollment.
13. Participants should have adequate organ function to be able to safely receive the approved standard of care regimens per the current FDA approved package insert, treating investigators discretion and institutional guidelines.
14. For females of reproductive potential: Negative urine and serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, serum pregnancy test will be required. Participants should be willing to use an adequate method of contraception for the course of the study through 120 days after last dose of study medication or through 180 days after last dose of chemotherapeutic agents. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
15. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks prior to administration of study regimen.
2. Has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
3. Has clinically active diverticulitis, intra-abdominal abscess, GI obstruction, abdominal carcinomatosis.
4. Prior treatment or history of allergy/hypersensitivity with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, or other specific T-cell co-stimulation or checkpoint targeting drugs.
5. Has a known sensitivity to any component of cisplatin, carboplatin, paclitaxel or pemetrexed
6. Participants with carcinomatous meningitis
7. Participants with active or suspected autoimmune diseases are excluded, with the following exceptions allowed: vitiligo, well-controlled type I diabetes mellitus, residual hypothyroidism due to autoimmune condition requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
8. Individuals who have received systemic corticosteroids or other immunosuppressive medications within the last 14 days prior to enrollment are excluded. Exceptions are made for topical, inhaled, nasal, ophthalmic steroids, or systemic corticosteroids at physiological doses not to exceed 10 mg/day of prednisone or an equivalent corticosteroid.
9. Participants with a history of ILD, or those who are suspected of having symptomatic ILD, or those with pneumonitis.
10. Individuals with a positive test for HIV, Hep B or Hep C are excluded unless it is well-controlled with no increased risk of immunosuppression and with no potential drug interactions with current antiviral therapy.
11. Participants with a history of other malignancies are excluded, except for those with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, or any cancer in situ that has been treated curatively, and the participant has been in complete remission for more than two years with any cancer prior to the start of the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-04-27 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Molecular Response in Patients with PD-L1 Negative Advanced NSCLC Treated with Dual vs. Single ICB Plus CT Regimens | Baseline to 64 days (C4D1)
  To assess and quantify the rate of molecular response, defined as the complete disappearance of circulating tumor DNA (ctDNA) from baseline levels, by Cycle 4 Day 1 (C4D1). This study compares patients with PD-L1 negative advanced non-small cell lung cancer (NSCLC) who are treated with a dual immune checkpoint blockade (ICB) plus chemotherapy (CT) strategy against those receiving a single ICB plus CT regimen. The objective explores whether the addition of a second ICB enhances the molecular response when integrated into standard chemoimmunotherapy protocols in this specific patient population.

SECONDARY OUTCOMES:
Efficacy Evaluation | Baseline up to 24 months
  To determine the Overall Response Rate (ORR) in patients receiving dual immune checkpoint blockade (ICB) plus chemotherapy (CT) and those receiving single ICB plus CT. The ORR will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Correlation Analysis | Baseline up to 24 months
  To investigate the correlation between ctDNA responses at Cycle 4 Day 1 (C4D1) and traditional RECIST v1.1 criteria in patients receiving dual versus single ICB plus CT. The analysis aims to validate ctDNA as a predictive biomarker for treatment response.

OTHER OUTCOMES:
Progression-Free Survival (PFS) | Baseline to 24 months
  To evaluate the median Progression-Free Survival (PFS) among patients treated with dual immune checkpoint blockade (ICB) plus chemotherapy (CT) compared to those receiving single ICB plus CT. The aim is to evaluate the impact of the combined treatment strategy on disease progression.
Median Overall Survival (OS) | Baseline to 24 months
  To evaluates the median Overall Survival (OS) in patients receiving dual ICB plus CT versus those treated with single ICB plus CT, offering insights into the long-term benefits of these treatment regimens.
Tolerability Assessment | Baseline to 24 months
  To assess the tolerability of dual versus single ICB plus CT strategies using patient-reported outcomes (PROs). The focus is on evaluating the patient experience and side effect profiles associated with these treatment options in patients with PD-L1 negative advanced NSCLC.

CONTACTS AND LOCATIONS:
Overall Officials: Aakash Desai, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States